CLINICAL TRIAL: NCT03839277
Title: Adenoma Detection Rate Using Endocuff Vision in China
Acronym: SinoEVADR
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: One investigator is out-of-service due to carrying out another task.
Sponsor: Changhai Hospital (Other)
Collaborators: Sixth Affiliated Hospital, Sun Yat-sen University (Other); Shanghai Zhongshan Hospital (Other); Tianjin People's Hospital (Other); Tianjin Nankai Hospital (Other)
Responsible Party: Principal Investigator, En-Da Yu, Director of Department of Colorectal Surgery and Vice Director of GI Endoscopy, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SINOCOLO2019A
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Colorectal Neoplasms; Colonic Polyp; Adenoma
Keywords: adenoma detection rate
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps; Adenoma

STUDY DESIGN:
Intervention Model Description: Endocuff Vision is a new device made of soft plastic material with a unique dynamic shape. It is manufactured by ARC Medical Design Limited and Diagmed in the United Kingdom. It has European Conformity in United Kingdom. The core is made of polypropylene and the 'finger like' projections are made of a thermoplastic elastomer. It comes in four colour coded sizes (purple, blue, green and orange) to fit a range of paediatric and adult colonoscopes. Endocuff Vision is the more updated version of device that has only one proximal row of more rounded finger-like projections. It is mounted at the tip of the colonoscope and held on by friction (pull-off force is a minimum of 10 Newtons).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endocuff Vision-assisted Colonoscopy (Active Comparator): Participants in this arm undergo Endocuff Vision-assisted colonoscopy
  Interventions: Device: Endocuff Vision
- Standard Colonoscopy (No Intervention): Participants in this arm undergo standard colonoscopy

INTERVENTIONS:
Device: Endocuff Vision — Endocuff Vision is attached to the tip of colonoscope before intubation.
  Arms: Endocuff Vision-assisted Colonoscopy

SUMMARY:
The primary aim of this study is

- to explore the usefulness of Endocuff Vision in colonoscopy on adenoma detection rate (ADR).

Other aims include to explore the data below when Endocuff Vision is used.

Mean adenomas detected per procedure, MAP Proximal Adenoma detection rate, pADR Polyp detection rate, PDR Proximal polyp detection rate, pPDR Mean polyps detected per procedure, MPP Withdrawal time, WT Cecal intubation rate, CIR Cecal intubation time, CIT

DETAILED DESCRIPTION:
Colorectal cancer is common in China. Most colorectal cancers happen when an adenoma becomes cancerous. Doctors use colonoscopy to look inside the colon and rectum and find adenomas and remove them. Removing adenomas is known to reduce the chances of a person developing colorectal cancers. The ability of colonoscopists finding adenomas varies, and there is a lot of researches into how to improve "adenoma detection rates".

A new device, called the Endocuff Vision has been shown to improve the rate of polyp detection at colonoscopy, and to make polyp removal easier. Previous studies have shown that there is a significant improvement in detection of adenomas when an Endocuff Vision is used (with the rate of detection of adenomas rising from 49% to 66%). Colonoscopists who have used the Endocuff Vision before also feel that polyp removal is easier when it is on the colonoscope. This study will randomise patients coming for colonoscopy to have their procedure performed as usual or as an Endocuff Vision-assisted colonoscopy. The investigators will record polyp and adenoma detection rates, duration of procedure, participant comfort levels, and complications. All patients referred for colonoscopy will be invited in 5 centres, recruiting a total of 1200 participants.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred for screening, surveillance, or diagnostic colonoscopy
* All patients must be able to give informed consent

Exclusion Criteria:

* Patients with any absolute contraindications to colonoscopy
* Patients with established or suspicion of large bowel obstruction or pseudo-obstruction
* Patients with known colon cancer or polyposis syndromes
* Patients with known colonic strictures
* Patients with known severe diverticular segments (that is likely to impede colonoscope passage)
* Patients with active colitis (ulcerative colitis, Crohn's colitis, diverticulitis, infective colitis)
* Patients lacking capacity to give informed consent
* Pregnancy
* Patients who are on clopidogrel, warfarin, or other new generation anticoagulants who have not stopped this for the procedure.
* Patients who are attending for a therapeutic procedure or assessment of a known lesion

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2019-06-12 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Adenoma detection rate, ADR | At the end of the procedure, up to 1 hour.
  ADR refer to the rate of adenoma detection, calculated as the proportion of subjects with at least one adenoma.

SECONDARY OUTCOMES:
Polyp detection rate, PDR | At the end of the procedure, up to 1 hour.
  PDR refer to the rate of polyp detection, calculated as the proportion of subjects with at least one polyp.

CONTACTS AND LOCATIONS:
Overall Officials: En-Da YU, Principal Investigator — Changhai Hospital
Locations (5):
- China (5):
  - Sixth affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Changhai Hospital, Shanghai, Shanghai Municipality
  - Tianjin Nankai Hospital, Tianjin, Tianjin Municipality
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ngu WS, Bevan R, Tsiamoulos ZP, Bassett P, Hoare Z, Rutter MD, Clifford G, Totton N, Lee TJ, Ramadas A, Silcock JG, Painter J, Neilson LJ, Saunders BP, Rees CJ. Improved adenoma detection with Endocuff Vision: the ADENOMA randomised controlled trial. Gut. 2019 Feb;68(2):280-288. doi: 10.1136/gutjnl-2017-314889. Epub 2018 Jan 23. PMID 29363535
- See also: PubMed link — http://www.ncbi.nlm.nih.gov/pubmed/29363535